CLINICAL TRIAL: NCT04627961
Title: A Phase 2 Trial of TAS 102 in Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: A Trial of LONSURF in Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP01/05/19
Record Dates: First submitted 2020-09-08; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Metastatic Nasopharyngeal Carcinoma; Recurrent Nasopharyngeal Carcinoma
Keywords: TAS102; NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Eligible patients who consent to participate will receive oral TAS-102 for days 1-5 and 8-12 of a 28 day cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): Patients with EBER positive nasopharyngeal carcinoma with recurrent or metastatic disease
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102 — Eligible patients who consent to participate will receive oral TAS-102 bid for days 1-5 and 8-12 of a 28 day cycle.
  Other Names: LONSURF

SUMMARY:
This is a single-arm, non-randomised study including patients with EBER positive nasopharyngeal carcinoma with recurrent or metastatic disease not amenable to curative treatment, who have received at least 1 regimen of platinum containing chemotherapy.

DETAILED DESCRIPTION:
HYPOTHESIS

Given the favourable activity of fluoropyrimidines (5Fluorouracil) which inhibit thymidylate synthase (TS) in nasopharyngeal carcinoma, the investigators hypothesized that TAS-102 may demonstrate efficacy in NPC through targeting TS as well as an additional mechanism of incorporating trifluridine triphosphate into DNA.

OBJECTIVES OF TRIAL

1. To determine the clinical efficacy of TAS-102 in recurrent and metastatic NPC
2. To assess the safety and tolerability of TAS-102 in the study population of R/M NPC
3. To study the pharmacokinetics of TAS-102 in the study population of R/M NPC
4. To study potential predictive biomarkers for clinical benefit from TAS-102

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written consent for the trial.
2. Participants who are at least 21 years of age on the day of signing informed consent with histologically or cytologically confirmed diagnosis of non-keratinizing nasopharyngeal carcinoma (NPC) that has recurred at loco regional and/or distant sites will be enrolled in this study.
3. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Have EBV-positive NPC by EBV-encoded small RNA in situ hybridization (EBER in situ hybridization [ISH]) assay. If EBV-positive status has been previously determined by EBER ISH assay, then no re-testing is required.

   Note: If EBV status by EBER ISH assay has not been previously determined, tumor tissue from archival tissue may be submitted for EBV determination.
5. Received one or more lines of chemotherapy, which must include prior treatment with a platinum agent and must not be amenable to potentially curative radiotherapy or surgery.
6. Willingness to donate blood for translational research studies.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Have an adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.

   Table 1 Adequate Organ Function Laboratory Values System Laboratory Value
   * Hematological

     1. Absolute neutrophil count (ANC) > 1.5x109/L
     2. Platelets ≥ 100 x109/L
     3. Hemoglobin ≥ 8.0 g/dL a
   * Renal

     a) Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥ 30 mL/min for participants with creatinine levels > 1.5X ULN
   * Hepatic

     1. Serum total bilirubin (Tbil) < 1.5 X ULN EXCEPT Patients with Gilbert's Syndrome, who can have Tbil < 3.0 mg/dL
     2. AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Coagulation

     1. International Normalized Ratio (INR) OR prothrombin time (PT) ≤ 1.5X ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
     2. Activated partial thromboplastin time (aPTT) ≤ 1.5X ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.
9. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study medication.
10. A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.

   Note: Participants must have recovered from all AEs to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible.

   Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
2. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
3. Has a known history of active TB (Bacillus Tuberculosis).
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
5. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast or cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.
6. Has known brain metastases or leptomeningeal metastases, whether treated or untreated. NOTE: Primary nasopharyngeal cancers that directly invade the skull base and extend into the infratemporal fossa (e) are not regarded as brain metastases and are not excluded.
7. Has an active infection requiring systemic therapy.
8. Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
12. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization/allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 45 months
  As defined by complete response (CR) + partial response (PR) + stable disease (SD) at 12 weeks of assessment using RECIST 1.1.

SECONDARY OUTCOMES:
Progression free survival rate of patients | 45 months
  as defined as the time from initiation of treatment to radiological progression, clinical deterioration or death.
Best objective response rate | 45 months
  as assessed by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] An X, Wang FH, Ding PR, Deng L, Jiang WQ, Zhang L, Shao JY, Li YH. Plasma Epstein-Barr virus DNA level strongly predicts survival in metastatic/recurrent nasopharyngeal carcinoma treated with palliative chemotherapy. Cancer. 2011 Aug 15;117(16):3750-7. doi: 10.1002/cncr.25932. Epub 2011 Feb 11. PMID 21319149
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774